CLINICAL TRIAL: NCT03526575
Title: Operational Ground Testing Protocol to Optimize Astronaut Sleep Medication Efficacy and Individual Effects
Brief Title: Optimize Astronaut Sleep Medication Efficacy and Individual Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0925-0586
Record Dates: First submitted 2018-03-26; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Sleep; Cognition; Pharmacologic Actions
MeSH Terms: interventions — Zolpidem; zaleplon

STUDY DESIGN:
Intervention Model Description: Experiment 1 will involve N=14 subjects randomized to placebo , 10 mg Zolpidem (Ambien) and 10 mg Zaleplon (Sonata) in counterbalanced order and will be awakened 90 min. post-placebo administration (half at 60 min and half at 90 min). The latter will be done to maintain some degree of blinding relative to the participants knowledge of conditions and the staff working on the protocol. Females and those subjects who have had a previous adverse experience with 10 mg zolpidem will be placed into Experiment 2, which will involve N=20 subjects randomized to placebo , 5 mg zolpidem and 10 mg zaleplon. Experiment 1 and 2 will provide data on zaleplon 10 mg compared to placebo on a total of 34 subjects consisting of astronauts and other subjects considered analogous to the astronaut population, which will provide the larger sample needed to identify those subjects who have cognitive performance deficits on abrupt awakening to the less sedating 10 mg zaleplon.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10 mg Zolpidem and 10 mg Zaleplon (Placebo Comparator): Experiment 1 will involve N= 14 subjects randomized to placebo , 10 mg zolpidem for males and 10 mg zaleplon in counterbalanced order. Subjects are nested into group.
  Interventions: Drug: Zolpidem
- 5 mg Zolpidem and 10 mg Zaleplon (Placebo Comparator): Experiment 2, which will involve N=20 subjects randomized to placebo, 5 mg zolpidem and 10 mg zaleplon. All females will be placed in experiment 2. Subjects are nested into group.
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem
  Other Names: Zaleplon

SUMMARY:
In the study titled Operational Ground Testing Protocol to Optimize Astronaut Sleep Medication Efficacy and Individual Effects (Phase 11), two randomized , blinded , placebo-controlled , cross-over trials will be conducted. The hypnotic medication and the placebo will be indistinguishable by subjects. Experiment 1 will involve N=14 subjects randomized to placebo , 10 mg Zolpidem (Ambien) and 10 mg Zaleplon (Sonata) in counterbalanced order and will be awakened 90 min. post-placebo administration (half at 60 min and half at 90 min). The latter will be done to maintain some degree of blinding relative to the participants knowledge of conditions and the staff working on the protocol. Zolpidem is the most commonly , and Zaleplon is the second most commonly , used sleep aid medication used in spaceflight. Females and those subjects who have had a previous adverse experience with 10 mg zolpidem will be placed into Experiment 2, which will involve N=20 subjects randomized to placebo , 5 mg zolpidem and 10 mg zaleplon. Data acquisition for both experiments will occur in the Astronaut Quarantine Facility ("AQF") at Johnson Space Center (JSC). Experimental methods and cognitive outcomes will be the same as those used in the pilot investigation titled Develop and Implement Operational Ground Testing Protocols to Individualize Astronaut Sleep Medication Efficacy and Individual Effects (Phase I). Combined , Experiment 1 and 2 will provide data on zaleplon 10 mg compared to placebo on a total of 34 subjects consisting of astronauts and other subjects considered analogous to the astronaut population (e.g., Flight Controllers, Flight Directors , Flight Surgeons, medical residents and medical students on National Aeronautics and Space Administration (NASA) rotation, and NASA/contractor employed University of Texas Medical Branch physician's) , which will provide the larger sample needed to identify those subjects who have cognitive performance deficits on abrupt awakening to the less sedating 10 mg zaleplon.

DETAILED DESCRIPTION:
The NASA /JSC Behavioral Health and Performance (BHP) Element of Space Medicine Division , Human Research Program (HRP) is supporting a ground-based directed research study to evaluate the effects of sleep medications (relative to placebo) on astronaut and other populations analogous to the astronaut population (e.g., Flight Controllers, Flight Directors, Flight Surgeons, medical residents and medical students on NASA rotation , and NASA/contractor employed University of Texas Medical Branch physician's) cognitive performance after an abrupt awakening. The second objective of the study is to develop a protocol to select a sleep medication and dose that minimally affects an individual 's cognitive performance upon awakening. Following completion of the study , it is the intent of the BHP Element to work with Space Medicine in the transition of the data and protocol as "best practices " for medical operations provided by the Clinical Services Branch in the Space Medicine Division at the NASA Johnson Space Center.

The study aims to characterize the effects of the most commonly used sleep medications and dosages on performance after an unplanned awakening , while providing the foundation for future development of individualized protocols for sleep medication use during training and on-orbit for astronauts and analogous populations (e.g., Flight Controllers , Flight Directors , Flight Surgeons , medical residents and medical students on NASA rotation , and NASA/contractor employed University of Texas Medical Branch physician's). Findings from the study will also further inform BHP 's development of an education training program related to countermeasures for sleep loss, circadian desynchronization , fatigue, and work overload for astronauts as well as ground crews who work night shifts in support of missions. Results of the study will also inform the human system health and medical standards and requirements for future exploration missions.

The study protocol was successfully pilot tested in the study titled Develop and Implement Operational Ground Testing Protocols to Individualize Astronaut Sleep Medication Efficacy and Individual Effects (Phase I) with N=7 subjects (6 NASA flight surgeons and 1 BHP Operations professional) as subjects from March through June , 2009. The pilot study results supported the scientific feasibility of conducting a randomized , blinded , placebo controlled study of sleep medication effects on alarm-based awakenings. Preliminary analysis from the pilot study indicated differences in performance upon abrupt awakening between the sleep medication and placebo conditions. Thus, the pilot data also supported the likelihood of new scientific and clinical insights from the Phase II studies with astronauts and the additional analogous populations (e.g., Flight Controllers, Flight Directors, Flight Surgeons, medical residents and medical students on NASA rotation, and NASA/contractor employed University of Texas Medical Branch physician's) .

In the study titled Operational Ground Testing Protocol to Optimize Astronaut Sleep Medication Efficacy and Individual Effects (Phase 11), two randomized , blinded , placebo-controlled , cross-over trials will be conducted. The hypnotic medication and the placebo will be indistinguishable by subjects. Experiment 1 will involve N=14 subjects randomized to placebo , 10 mg Zolpidem (Ambien) and 10 mg Zaleplon (Sonata) in counterbalanced order and will be awakened 90 min. post-placebo administration (half at 60 min and half at 90 min). The latter will be done to maintain some degree of blinding relative to the participants knowledge of conditions and the staff working on the protocol. Zolpidem is the most commonly , and Zaleplon is the second most commonly , used sleep aid medication used in spaceflight. Females and those subjects who have had a previous adverse experience with 10 mg zolpidem will be placed into Experiment 2, which will involve N=20 subjects randomized to placebo , 5 mg zolpidem and 10 mg zaleplon. Data acquisition for both experiments will occur in the Astronaut Quarantine Facility ("AQF") at JSC. Experimental methods and cognitive outcomes will be the same as those used in the pilot investigation titled Develop and Implement Operational Ground Testing Protocols to Individualize Astronaut Sleep Medication Efficacy and Individual Effects (Phase I). Combined , Experiment 1 and 2 will provide data on zaleplon 10 mg compared to placebo on a total of 34 subjects consisting of astronauts and other subjects considered analogous to the astronaut population (e.g., Flight Controllers, Flight Directors , Flight Surgeons, medical residents and medical students on NASA rotation, and NASA/contractor employed University of Texas Medical Branch physician's) , which will provide the larger sample needed to identify those subjects who have cognitive performance deficits on abrupt awakening to the less sedating 10 mg zaleplon.

This is an applied study and it is not feasible to include two or three doses of each drug in order to determine a dose-response curve based on each of the drugs pharmacodynamics. Literature has shown that zaleplon 10 mg will be less disruptive on performance at awakening than zolpidem 10 mg and that zaleplon 20 mg is likely to be comparable in effects to zolpidem 10 mg. However , zaleplon 20 mg is not a commonly used dose in space, whereas zolpidem 10 mg and 5mg, and zaleplon 10 mg are used-hence the study will focus on these drugs and doses. More importantly , the goal of this study is not to determine whether these dose-by-drug comparisons are likely to yield the same average results in astronauts as has been found in the general population (e.g., Roehrs et a., 1994; Wesensten et al., 1996; Greenblatt et al., 1998; Hindmarch et al., 2001). Instead , we began by are focusing on individual astronaut vulnerability to hypnotic sedation on awakening , and having a limited number of astronauts who can realistically participate in the operational research was not realistic or conducive in completing the study. We needed to expand our astronaut population to include international astronauts and other populations deemed analogous to the astronaut population (e.g., Flight Controllers, Flight Directors , Flight Surgeons, medical residents and medical students on NASA rotation,and NASA/contractor employed University of Texas Medical Branch physician's) . We want to evaluate as many astronauts on these drugs and doses as possible , and in a manner that permits comparisons between both drug type and dose; however , it became necessary to broaden our subject pool in order to reach the desired N. Thus Experiment 1 will evaluate 10 mg zolpidem for males and zaleplon 10 mg relative to placebo in N=14 astronauts and analogous subjects (e.g., Flight Controllers, Flight Directors, Flight Surgeons, medical residents and medical students on NASA rotation,and NASA/contractor employed University of Texas Medical Branch physician's). Experiment 2 will evaluate zolpidem 5 mg and zaleplon 10 mg relative to placebo in N = 20 additional astronauts and other analogous subjects (e.g., Flight Controllers , Flight Directors , Flight Surgeons, medical residents and medical students on NASA rotation,and NASA/contractor employed University of Texas Medical Branch physician's).

ELIGIBILITY:
Inclusion Criteria:

The participant must be an active astronaut or analogous to the astronaut population (e.g., Flight Controllers, Flight Directors, Flight Surgeons, medical residents and medical students on NASA rotation, and NASA /contractor employed University of Texas Medical Branch physician's) to participate in the study. Not Applicable (NA)

Exclusion Criteria:

Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Number of lapses of attention | 3 weeks
  The number of lapses of attention on 3 minute Psychomotor Vigilance Test

SECONDARY OUTCOMES:
Digit Symbol Substitution Test | 3 weeks
  The number of correct responses
Descending Subtraction Test | 3 weeks
  The number of correct responses
Free Recall | 3 weeks
  The number of correctly recalled words
Response time to shut off alarm time | 3 weeks
  The time subjects require to shut off the awakening simulated International Space Station (ISS) alarm

CONTACTS AND LOCATIONS:
Overall Officials: Smith Johnston, MD, Principal Investigator — JSC NASA; David Dinges, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dinges DF, Basner M, Ecker AJ, Baskin P, Johnston SL. Effects of zolpidem and zaleplon on cognitive performance after emergent morning awakenings at Tmax: a randomized placebo-controlled trial. Sleep. 2019 Mar 1;42(3):zsy258. doi: 10.1093/sleep/zsy258. PMID 30576525